CLINICAL TRIAL: NCT06523400
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Investigate the Efficacy and Safety of Once Daily Mexiletine PR During 26 Weeks of Treatment in Patients With Myotonic Dystrophy Type 1 and Type 2 (Phase 3)
Brief Title: The Efficacy and Safety of Once Daily Mexiletine PR in Patients With Myotonic Dystrophy Type 1 and Type 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Collaborators: Lupin Atlantis Holdings S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEX-DM-302
Record Dates: First submitted 2024-05-03; First posted 2024-07-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, parallel-group, placebo-controlled study intended to evaluate the efficacy and the safety of mexiletine PR in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2). The study will consist of a 4-week screening period and a 26-week treatment phase with patient visits at screening, baseline, Weeks 1, 2, 14, and 26. Eligible patients will be randomized to mexiletine or placebo in a 1:1 ratio. Approximately 80 DM1 patients (40 active: 40 placebo) are planned to be enrolled. For the purpose of sample size re-estimation, an interim analysis will be conducted when a total of 40 patients complete/early terminate the study. In addition, 16 DM2 patients are planned to be enrolled (sub-group - 8 active: 8 placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mg (matching sachet volumes to low, medium and high dose active drug)
  Interventions: Drug: Placebo
- Mexiletine prolonged-release (PR) (Active Comparator): Mexiletine PR 167 mg (mexiletine HCl 200 mg) Mexiletine PR 333 mg (mexiletine HCl 400 mg) OR Mexiletine PR 500 mg (mexiletine HCl 600 mg)
  Interventions: Drug: Mexiletine granules for prolonged-release oral suspension

INTERVENTIONS:
Drug: Mexiletine granules for prolonged-release oral suspension — Mexiletine PR
  Arms: Mexiletine prolonged-release (PR)
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-Controlled, Multi-Center Study to Investigate the Efficacy and Safety of Once Daily Mexiletine PR During 26 Weeks of Treatment in Patients with Myotonic Dystrophy Type 1 and Type 2 (HERCULES study)

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study intended to evaluate the efficacy and the safety of mexiletine PR in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2). The study will consist of a 4- week screening period and a 26-week treatment phase with patient visits at screening, baseline, Weeks 1, 2, 14, and 26. Eligible patients will be randomized to mexiletine or placebo in a 1:1 ratio. Approximately 80 DM1 patients (40 active: 40 placebo) are planned to be enrolled. For the purpose of sample size re-estimation, an interim analysis will be conducted when a total of 40 patients in total complete/early terminate the study.

In addition, 16 DM2 patients are planned to be enrolled (sub-group - 8 active: 8 placebo).

ELIGIBILITY:
Inclusion Criteria:

1. DM1 or DM2 diagnosis confirmed genetically;
2. Ability to comprehend and willingness to sign an informed consent (ICF) or ICF of the parent(s)/legal guardian and written assent from the patient (if patient < 18 years of age);
3. Ability to understand the study requirements including intention to stay in the study until the end-of-study visit at 26 weeks of treatment;
4. Male or non-pregnant female ≥16 years of age;
5. Body Mass Index (BMI) of 18.5 kg/m2 to 30 kg/m2, and weight ≥45 kg;
6. Female patients of childbearing potential must be using a highly effective form of birth control for the duration of the study and for at least 7 days after last dose of study drug;
7. No significant cardiac abnormalities as determined by a cardiologist's assessment;
8. Have sufficient finger flexor strength to grasp the handle of the dynamometer used to measure myotonia;
9. Presence of clinical handgrip myotonia (delayed relaxation of grip of ≥ 3 seconds after maximum voluntary contraction) at screening using VHOT;
10. Be able to walk independently 10 meters (cane, walker, orthoses allowed);
11. DM1 patients only - Muscular impairment rating scale (MIRS) score of 2, 3 or 4.-

Exclusion Criteria:

1. Are pregnant or lactating;
2. Have any one of the following medical conditions: uncontrolled diabetes mellitus, cancer other than skin cancer less than five years previously (e.g., basal-cell carcinoma (BCC) and squamous-cell carcinoma (SCC) of skin allowed), multiple sclerosis, seizure disorders, or other serious medical illness;
3. Severe renal impairment (glomerular filtration rate (GFR) < 30 mL/min);
4. Medical conditions which could interfere with muscle function such as infections, trauma, fractures, or planned surgery;
5. Medical conditions that could affect hand functioning including but not limited to rheumatoid arthritis, Dupuytren's contracture, hand deformity, etc.;
6. Severe arthritis or medical condition (other thanDM1/DM2) that would significantly impact ambulation;
7. High incidence of falls or fall-associated fractures (>5 falls during the past 12 months);
8. Preexisting elevated liver function tests > 3 times the upper limit of normal (ULN) at screening (alanine transaminase (ALT)/aspartate transaminase (AST), gamma-glutamyl transferase (GGT)) and/or any abnormal chemistry, hematology or urine lab considered clinically significant by investigator;
9. Serum potassium values < 3.5 mmol/L or > 5.0 mmol/L or serum magnesium values < 1.7 mg/dL. Electrolytic imbalance such as hypokalaemia, hyperkalaemia or hypomagnesaemia may increase the proarrhythmic effects of mexiletine. Electrolyte imbalances need to be corrected before administering mexiletine and will be monitored throughout treatment.
10. Treatment with mexiletine within 4 weeks prior to baseline (Day 1);
11. Intake of any anti-myotonic treatment within 4 weeks prior to baseline (Day 1) or 5 half-lives, whichever is longer such as metformin, such as propafenone, flecainide, lamotrigine, carbamazepine or any other channel-blocker/ anticonvulsive drugs;
12. Use of any concomitant medications that could increase the cardiac risk;
13. Known allergy to mexiletine or any local anesthetics;
14. Participation in another interventional clinical study during the last 3 months or 5 half-lives of the investigational medicinal product, whichever is longer;
15. Wheelchair-bound or bed-ridden;
16. Any cardiac safety associated condition including any of the following criteria detected by screening cardiac evaluations including 24-hr Holter monitor, echocardiogram and clinical evaluations:

    * PR interval ≥240 ms or QRS duration ≥120 ms on resting ECG
    * Personal history of 3rd degree or 2nd degree type 2 atrioventricular block or sinus node dysfunction with pauses ≥3 seconds, complete bundle branch block, bifascicular and trifascicular block or any heart block susceptible to evolve to complete heart block
    * Personal history of sustained atrial fibrillation, flutter or tachycardia (duration >30 seconds)
    * Personal history of non-sustained (ventricular triplets or more) or sustained ventricular tachycardia
    * Myocardial infarction (acute or past) or coronary artery stenosis >50%, presence of abnormal Q waves
    * New York Heart Association (NYHA) Class II to IV heart failure
    * Left ventricular systolic dysfunction with ejection fraction <50%
    * Sinus node dysfunction (including ECG sinus rate <50 beats per minute (BPM))
    * Co-administration of antiarrhythmics inducing torsades de pointes (class Ia: quinidine, procainamide, disopyramide, ajmaline; class Ic: encainide, flecainide, propafenone, moricizine; class III: amiodarone, sotalol, ibutilide, dofetilide, dronedarone, vernakalant)
    * Co-administration of other classes of antiarrhythmics (class Ib: lidocaine, phenytoin, tocainide; class II: propranolol, esmolol, timolol, metoprolol, atenolol, carvedilol, bisoprolol, nebivolol; class IV: verapamil, diltiazem)
    * Patients with implantable cardioverter defibrillators (ICDs) and pacemakers are excluded
    * Presence of symptomatic coronary artery disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of once daily mexiletine PR for the symptomatic treatment of myotonia in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2). | 26 weeks
  Handgrip relaxation time in DM1 patients by mean change in baseline of handgrip relaxation time (seconds) after maximal voluntary isometric contraction (MVIC)

SECONDARY OUTCOMES:
To assess the safety of once daily mexiletine PR for the symptomatic treatment of myotonia in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2). | 26 weeks
  Number and frequency of AEs/SAEs throughout the study while on treatment
Mean change in VAS | 26 weeks
  Score for muscle stiffness (myotonia severity) as self-reported by patients on a Visual Analog Scale (VAS)
Mean change in MBS scores | 26 weeks
  Mean change in Myotonia Behavior Scale (MBS) scores
Mean change in health-related quality of life | 26 weeks
  Mean change in health-related quality of life (measured by INQoL)
Mean change in DM1-Activ-c scale (DM1 patients only) | 26 weeks
  Mean change in measure of activity and social participation (measured by a Rasch-built scale with a 0-100 interval range)
Mean change in time to perform the 10-meter Walk Test | 26 weeks
  Mean change in time (seconds) to perform the 10-meter Walk Test (10mWT)
Mean change in handgrip relaxation time | 26 weeks
  Mean change in maximal voluntary isometric contraction (MVIC) and relaxation time by Video-recording of Hand Opening Time (VHOT) functional evaluation
Mean change in time to perform Timed-up and go (TUG) test | 26 Weeks
  Mean change in time (seconds) to perform Timed-up and go (TUG) test
Mean change in health-related quality of life measured by EQ-5D | 26 weeks
  Mean change in health-related quality of life measured by EQ-5D (5-point scale)
Mean change in Myotonic Dystrophy Health Index (MDHI) score (DM1 patients) | 26 weeks
  Mean change in Myotonic Dystrophy Health Index (MDHI) score (DM1 patients) as measured by patient's perceived health
Mean change in Myotonic Dystrophy 2 Health Index (MD2HI) score (DM2 patients) | 26 weeks
  Mean change in Myotonic Dystrophy 2 Health Index (MDHI) score (DM2 patients) as measured by patient's perceived health
Assess the safety of mexiletine PR by changes in ECG | 26 weeks
  Mean change in ECG (PR, QRS, QTc intervals, average HR) from baseline
Assess the safety of mexiletine PR by AEs | 26 weeks
  Incidence of treatment emergent adverse events (TEAEs), treatment-related TEAEs, serious AEs, and patient discontinuation rate
Assess the safety of mexiletine PR by standard clinical laboratory evaluations | 26 weeks
  Assess the safety of mexiletine PR by standard clinical laboratory evaluations as measured by hematology, chemistry, and urinalysis assessments from change in baseline
Assess the safety of mexiletine PR by vital signs | 26 weeks
  Assess the safety of mexiletine PR by vital signs (pulse, respiration, body temperature, and blood pressure) from change in baseline
Assess the safety of mexiletine PR by physical examinations | 26 weeks
  Assess the safety of mexiletine PR by change in baseline from physical examinations
To assess the pharmacokinetics of mexiletine PR | 26 weeks
  To assess the pharmacokinetics of mexiletine PR as measured by PK parameter AUC0-t
To assess the pharmacokinetics of mexiletine PR by AUC0-t | 26 weeks
  To assess the pharmacokinetics of mexiletine PR as measured by PK parameter AUC0-t (area under the concentration-time curve from time zero to last timepoint)
To assess the pharmacokinetics of mexiletine PR by Cmax | 26 weeks
  To assess the pharmacokinetics of mexiletine PR as measured by PK parameter Cmax (maximum plasma concentration)

CONTACTS AND LOCATIONS:
Locations (7):
- Laboratory for Muscle Diseases and Neuropathies, Leuven, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- Ludug-Maximilians University, München, Germany
- Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Italy
- University Hospital of Madrid, Madrid, Spain
- United Kingdom (2):
  - Saint George's University Hospitals NHS Foundation Trust, London
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No